CLINICAL TRIAL: NCT03972826
Title: Epicenters for the Prevention of Healthcare Associated Infections (HAIs) -- Volume of Contamination and Nosocomial Infection Control: Specific Aim II.1
Brief Title: Use of Provodine to Protect HCW Hands (Aim II.1)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Supplier of product went into bankruptcy proceedings
Sponsor: University of Iowa (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Microdermis Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1U54CK000448-01 (NIH)
Record Dates: First submitted 2019-05-29; First posted 2019-06-04 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Infection
Keywords: hand hygiene; healthcare worker self-contamination
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Other): Subjects serve as self-controls. Subjects first perform hand-hygiene with alcohol-based hand rub then doff gloves contaminated with either S. marcescens or MS2 phage and the hands are cultured using a bag-broth method to determine whether the subjects self-contaminated while doffing. Subjects then clean their hands thoroughly, perform hand hygiene with Provodine, then repeat the doffing and culture process.
  Interventions: Other: Provodine

INTERVENTIONS:
Other: Provodine — Subjects serve as self-controls. Subjects first perform hand-hygiene with alcohol-based hand rub then doff gloves contaminated with either S. marcescens or MS2 phage and the hands are cultured using a bag-broth method to determine whether the subjects self-contaminated while doffing. Subjects then clean their hands thoroughly, perform hand hygiene with Provodine, then repeat the doffing and culture process.

SUMMARY:
The investigators will assess whether applying Provodine, an FDA-approved hand hygiene product with a long duration of anti-microbial action, to healthcare workers' hands protects against self-contamination during the removal of personal protective equipment (gloves, gowns, etc).

DETAILED DESCRIPTION:
We will perform a two-armed pilot test among 40 front-line healthcare workers (nurses, doctors, respiratory therapists, etc) at the University of Iowa Hospitals and Clinics. Participants will serve as their own controls. First, participants will perform hand hygiene with alcohol-based hand rub as they normally would in clinical practice then don PPE. We, the research team, will contaminate participating healthcare workers' (HCW) PPE with either bacteriophage MS2 (twenty participants) or S. marcescens ATCC 14756 (twenty participants). MS2 preparation and propagation and S. marcescens culture suspensions will each be performed as previously described. The MS2 bacteriophage will be suspended in 0.01 M phosphate-buffered saline and each PPE site will be contaminated with 10^5 plaque-forming units (PFU) of MS2 in 5 drops of 5 μL each. Aliquots of 3 mL of S. marcescens broth suspension (yielding bacterial titers of ~1 X 10^9 CFU/ml) will be applied to each PPE site. Participants will then doff PPE using the Centers for Disease Control's (CDC) recommended protocol. We will sample their hands using the bag broth method. A research assistant will monitor participants as they wash their hands with soap and water then rinse their hands with 70% ethanol. Participants will then apply ProvodineTM to their hands and put on (don) fresh PPE. We will repeat the contamination, doffing, and sampling procedure. For MS2 recovery, we will assay the eluent using the most probable number (MPN) enrichment infectivity assay. For S. marcescens recovery, we will dilute the eluent, plate it, incubate the plates, and count the colonies as described.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be UIHC healthcare workers (doctors, nurses, etc.)

Exclusion Criteria:

* Known skin sensitivity to povidone iodine or Provodine (TM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Percent of participants whose hands were colonized after doffing gloves | 30 minutes
  The percent of participants whose hands were contaminated with either S marcescens or the phage MS2 after doffing gloves when participants did hand hygiene before the trial with an alcohol-based hand rub compared with that when participants had done hand hygiene before the trial with Provodine
Colony-forming units (CFU) or Plaque forming units (PFU) on participants' hands | 30 minutes
  The number of S. marcescens CFU or MS2 plaque forming units (PFU) on participants hands when they did hand hygiene before the trial with an alcohol-based hand rub compared with when participants had done hand hygiene before the trial with Provodine

CONTACTS AND LOCATIONS:
Overall Officials: Loreen Herwaldt, MD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-10-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT03972826/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT03972826/ICF_001.pdf